CLINICAL TRIAL: NCT06157138
Title: Incidence of B-Lines in Pulmonary Echography, in Patients Undergoing Open Abdominal Surgery.
Brief Title: Observation of B-lines in Pulmonary Echography, During Open Abdominal Surgery
Acronym: LUS-SURG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Augusto Rolle, MD, MSc, Pontificia Universidad Catolica de Chile
Other Study IDs: 230209001
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Open Abdominal Surgery; Lung Ultrasound
Keywords: lung ultrasound; B-Lines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing open abdominal surgery: Patients older than 18 years undergoing open abdominal surgery. They will be followed by a protocol of pulmonary echography during and after surgery in the postoperative care unit

SUMMARY:
There is no a reliable marker of intraoperative fluid excess or overload. The use of lung ultrasound in other settings, such as emergency room and critical care patients, helps us to determine if a patient has a condition of augmented intrathoracic fluid, that could be related to several circumstances, such as fluid overload, but also to heart failure, in example.

Nevertheless, there is no information regarding the basal incidence of this finding, to ascertain if could be eventually used as a potential marker of fluid overload. This protocol looks for the incidence of the finding of B-Lines, which are related to fluid overload, in patients undergoing open abdominal surgery.

DETAILED DESCRIPTION:
The presence of B-lines will be observed in 4 spaces at each evaluation: Anterior-superior, and infero-lateral, by each side.

The times of evaluation will be prior to intubation, after intubation, every one hour of surgery, at the end of the surgery prior to extubation, and after 2 hours in the postoperative care unit.

Other variables addressed will be the vital signs, parameters related to a diminished intravascular status (ie, pulse pressure variability), central venous pressure, volume changes (reposition, bleeding, diuresis), and requirements of blood products.

A correlation with baseline characteristics of patients will be observed; nevertheless, this study is directed as primary endpoint to evaluate the incidence of the B-lines in echography, and the sample size was calculated following this endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to open abdominal surgery Older than 18 years.

Exclusion Criteria:

* Previous thoracic surgery, BMI over 30 kg/m2 Baseline respiratory alterations related to preoperative supplementary oxygen requirements Evident malformations of the thoracic wall If the position required for the surgery does not allow the echographic windows required for the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to open abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Apparition of pulmonary B-Lines | During surgery and after 2 hours in the postoperative care unit
  3 or more B-Lines in any evaluated quadrant

SECONDARY OUTCOMES:
Postoperative pulmonary complications | After 2 hours in the postoperative care unit
  Requirements of supplementary oxygen at PACU discharge or postoperative mechanical ventilatory support
fluid administration and B lines | During surgery
  Correlation of fluid administration and appearance of B lines

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Rolle, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico UC-Christus, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
Not required; all the data will be managed by the research team